CLINICAL TRIAL: NCT02411617
Title: Single vs. Double Drain in Modified Radical Mastectomy: A Randomized Control Trial
Brief Title: Single vs. Double Drain in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memon Medical Institute (Other)
Responsible Party: Principal Investigator, salma khan, Consultant General Surgeon, Memon Medical Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC:02
Record Dates: First submitted 2015-02-27; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single drain in modified radical mastectomy (Active Comparator): Post modified radical mastectomy with either one or two drains Intervention is use of single or double drain
  Interventions: Device: Drain
- Double drain in modified radical mastectomy (Active Comparator): Post modified radical mastectomy with either one or two drains Intervention is use of single or double drain
  Interventions: Device: Drain

INTERVENTIONS:
Device: Drain — Post modified radical mastectomy with either one or two drains Intervention is use of single or double drain

SUMMARY:
Seroma is a common complication following modified radical mastectomy(MRM). Closed drainage is used routinely to reduce incidence of seroma. Usually two drains are used in patients who underwent MRM to reduce post operative seroma. It is often associated with significant patient discomfort and prolonged fluid drainage.

The aim of this study is to evaluate effect of number of drains on seroma formation rate, postoperative pain and hospital stay during the immediate postoperative period after mastectomy for breast cancer.

DETAILED DESCRIPTION:
Modified Radical mastectomy is commonly performed procedure for carcinoma breast. After surgery two drains are placed, one in axilla and one beneath the flap. The use of two drains is associated with significant post operative discomfort and pain. On the other hand two drains have not been proven to decrease post operative seroma formation.

ELIGIBILITY:
Inclusion Criteria:

* All female patients underwent MRM for biopsy proven carcinoma breast

Exclusion Criteria:

* Immediate reconstruction
* Patient refusal to participate in study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
seroma formation | 30 days post surgery
  fluid collection beneath the flap sufficient to cause patient discomfort and pain

SECONDARY OUTCOMES:
Duration of hospital stay,, | 30 days after surgery
wound infection | 30 days after surgery
  as described by center of disease control (CDC) criteria
postoperative pain | 30 days after surgery
  measured on visual analogue scale (1 to 10) in first 24 hours after surgery.
hematoma | 30 days after surgery
  blood collection under the flap
flap necrosis | 30 days after surgery
  flap discoloration due to compromised blood supply of flap

REFERENCES:
- [Derived] Khan S, Khan M, Wasim A. Single vs. double drain in modified radical mastectomy: A randomized controlled trial. Turk J Surg. 2023 Jun 19;39(2):145-152. doi: 10.47717/turkjsurg.2023.5666. eCollection 2023 Jun. PMID 38026913